CLINICAL TRIAL: NCT02714894
Title: Glutamatergic System and Response to Clozapine in Patients With Treatment-Resistant Schizophrenia: a Prospective Proton Magnetic Resonance Spectroscopy Study
Brief Title: Response to Clozapine in Treatment Resistant Schizophrenia: A Longitudinal Magnetic Resonance Spectroscopy Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Ariel Graff, Ariel Graff MD, PhD, Centre for Addiction and Mental Health
Other Study IDs: 122-2015
Record Dates: First submitted 2016-03-14; First posted 2016-03-22 (Estimated); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Schizophrenia
Keywords: magnetic resonance imaging; magnetic resonance spectroscopy
MeSH Terms: conditions — Schizophrenia | interventions — Clozapine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Clozapine Responders (Non-URS): Definition of non-URS
  (1) ≥30% decrease in the PANSS positive subscale score, CGI-severity ≤3 and CGI-Improvement ≤2 after 12 weeks of treatment.
  Interventions: Drug: Clozapine
- Clozapine Non-Responders (URS): Definition of URS
  1. Taking clozapine for ≥ 12 weeks, attaining a plasma clozapine level ≥350 ng/ml.
  2. CGI-Severity score of ≥4 and score of ≥4 on 2 PANSS positivesymptom items.
  Interventions: Drug: Clozapine
- Healthy Controls: Healthy controls will be matched as closely as possible on age and gender with participants in the patient groups.

INTERVENTIONS:
Drug: Clozapine — Patient participants will be starting clozapine as part of their clinical care.
  Other Names: Clozaril
  Groups: Clozapine Non-Responders (URS); Clozapine Responders (Non-URS)

SUMMARY:
The purpose of this study is to investigate the relationship between glutamate and related brain chemicals and treatment response to clozapine in patients with treatment-resistant schizophrenia.

DETAILED DESCRIPTION:
This study will be a prospective proton spectroscopy (1H-MRS) study designed to compare the levels of glutamate, glutamine, glx, and glutathione in age- and gender- matched patients with poor response to clozapine (URS), patients with good response to clozapine (non-URS), and healthy controls. Participants with schizophrenia who fail to respond to optimal treatment with at least two different non-clozapine antipsychotics (i.e. treatment-resistant schizophrenia [TRS]) and who are starting clozapine as part of their clinical care will be recruited. A sample of healthy controls will also be recruited. Participants with TRS will have two 1H-MRS scans. The 1H-MRS scan will be performed within 1 week and 12 weeks after clozapine initiation. Clinical assessments will be performed within 1 week of each 1H-MRS scan and after 6 weeks of clozapine treatment. Cognitive assessments will also be performed within 1 week of 1H-MRS scans. Healthy controls will also undergo two 1H-MRS scans with a 12-week interval. Cognitive assessments will also be performed within 1 week of 1H-MRS scans.

ELIGIBILITY:
Inclusion Criteria for Participants with TRS:

* DSM-IV/SCID diagnosis of schizophrenia, schizoaffective disorder, delusional disorder, or psychotic disorder NOS.
* Age 18 years or older at time of scanning
* History of failure to respond to at least two previous sequential antipsychotic treatments different to clozapine, each attaining a chlorpromazine daily dose of≥ 400 mg for a duration ≥ 6 consecutive weeks.Long-acting antipsychotic treatment will not be allowed during the last trial prior to clozapine in order to avoid residual concentrations or effects.Failure of treatment will be defined by a Clinical Global Impression Severity (CGI-Severity) score of ≥4 and score of ≥4 on 2 Positive and Negative Syndrome Scale (PANSS) positive symptom items. The CGI-Severity or Global Assessment of Functioning (GAF) will be completed retrospectively based on information provided by the participant, participant's psychiatrist, medical chart, or other sources of available collateral information.

Exclusion Criteria for Participants with TRS:

* Incapacity to provide consent to participate in the research study.
* Substance abuse or dependence (within past six months), excluding nicotine and caffeine.
* Positive urine drug screen for drugs of abuse.
* Metal implants or a pace-maker that would preclude the MRI scan.
* History of head trauma resulting in loss of consciousness > 30 minutes that required medical attention.
* Unstable physical illness or significant neurological disorder including a seizure disorder.
* Size of head, neck, and body being unable to fit MRI scanners.
* Refusal to provide consent to investigator to communicate with physician of record to obtain collateral information.
* Psychiatric concerns raised by the physician of record regarding participation in the study.
* Currently taking medications that may directly impact the glutamatergic system (i.e. lamotrigine, topiramate, memantine or N-acetylcysteine)
* ECT, MST or TMS in the past 6 months

Inclusion criteria for Healthy Controls:

* Age of 18 and older at time of scanning
* Being capable to consent to study procedures
* Absence of history of psychiatric illness using the Mini-International Neuropsychiatric Interview (MINI)

Exclusion criteria for Healthy Controls:

* First degree family member with primary psychotic disorder
* Substance abuse or dependence (within past six months), excluding nicotine and caffeine.
* Positive urine drug screen for drugs of abuse
* Pacemakers, metallic cardiac valves, magnetic material such as surgical clips, implanted electronic infusion pumps or any other conditions that would preclude the MRI scan
* Clinically significant claustrophobia
* History of head trauma resulting in loss of consciousness > 30 minutes that required medical attention
* Size of head, neck, and body being unable to fit MRI scanners
* Unstable physical illness or significant neurological disorder including a seizure disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with schizophrenia who fail to respond to optimal treatment with at least two different non-clozapine antipsychotics (i.e. treatment-resistant schizophrenia [TRS]) and are starting clozapine will be recruited. A sample of healthy controls will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in 1H-MRS glutamatergic metabolites before and after clozapine. | Change from baseline (pre-clozapine) of 1H-MRS glutamatergic metabolites at 12 weeks
  1H-MRS will be employed to quantify glutamatergic metabolites, specifically glutamate, glutamine, glx and glutathione.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Graff, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world — http://www.camh.ca/en/research